CLINICAL TRIAL: NCT05235113
Title: Tele-exergame: Remotely-supervised Exercise Platform for Improving Cognition and Motor Function Using Telemedicine
Brief Title: Remote Game-based Exercise Program for Cognitive and Motor Function Improvement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: BioSensics (Industry); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Bijan Najafi, PhD, Professor of Surgery, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-1331; R44AG067909 (NIH)
Record Dates: First submitted 2021-11-05; First posted 2022-02-11 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Mild Cognitive Impairment; Dementia; Cognitive Impairment; Memory Loss
Keywords: tele-exercise; exergame; tele-rehabilitation; Telehealth; telemedicine; virtual reality
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Memory Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to intervention (IG) or control group (CG) with ratio of 1:1. The entire cohort will perform leg and foot exercises twice a week. The IG will use the Tele-exergaming platform, and the CG will do the exercises without the platform.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Remote Exercise with tele-exergame (Active Comparator): Subjects will perform exercises remotely twice a week with tele-exergaming platform.
  Interventions: Device: Tele-Exergame Platform
- home-based exercise without technology (Sham Comparator): Subjects will perform exercises at home without tele-exergaming platform twice a week.
  Interventions: Device: No Tele-Exergame Platform

INTERVENTIONS:
Device: Tele-Exergame Platform — Subjects will perform exercises remotely twice a week with tele-exergaming platform.
  Arms: Remote Exercise with tele-exergame
Device: No Tele-Exergame Platform — Subjects will perform exercises in the home exercise twice a week without tele-exergaming platform.
  Arms: home-based exercise without technology

SUMMARY:
As our population ages, more older adults face motor-cognitive declines, increasing their risk of falls and fear of falling. Exercise is an effective way to maintain cognitive function, as supported by recent studies. However, those with poor motor and cognitive abilities often struggle to visit rehabilitation centers, leading to high dropout rates and low adherence to unsupervised programs. A remote exercise program tailored for individuals with cognitive impairments is urgently needed to preserve cognitive function, promote independent living, and reduce related costs. Researchers aim to develop an in-home system for adults with mild cognitive issues or dementia, designed to improve balance and cognition while being remotely supervised through telemedicine.

DETAILED DESCRIPTION:
This study aims to develop and validate a remote exercise intervention for individuals at risk of or experiencing dementia using a wearable sensor-enabled platform, called Tele-Exergame. This approach could preserve cognitive function, promote independent living, reduce costs related to cognitive-motor decline, and advance remote technology use for screening cognitive and motor performance in older adults. The findings are crucial for healthcare providers, clinicians, seniors, and caregivers.

100 participants will be randomly assigned to either the intervention or control group, both undergoing a 12-week daily home exercise program for at least cumulative active exercise of 30 minutes per week twice weekly. The intervention group will complete sessions remotely using Tele-exergame, while the control group will participate in home-based exercise without technology.

ELIGIBILITY:
Inclusion Criteria:

* Adults with diagnosed with dementia or cognitive impairment
* Living independently in a residential home with a caregiver/informant
* Able to walk at least 30 feet with or without assistance

Exclusion Criteria:

* Immobility or major mobility disorder or inability to engage safely in the proposed weight-bearing exercise program
* Diagnosed with severe cognitive impairment (MoCA score < 16)
* Subjects with major hearing/visual impairment

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-11-03 (Actual); Primary Completion 2026-11-09 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Balance | Baseline and 12 weeks
  Change in balance from baseline to 12 weeks will be measured. Balance will be assessed by measuring center of mass sway. The investigator will use a validated wearable platform (BalanSen) to measure body sway.
Change in Cognitive Function | Baseline and 12 weeks
  Changes from baseline in cognitive function at 12 weeks. Cognitive performance will be assessed using Montreal Cognitive Assessment (MoCA). Scores on the MoCA range from zero to 30, with a score of 26 and higher generally considered normal.

SECONDARY OUTCOMES:
Change in Physical Activity | Baseline and 12 weeks
  Changes in physical activity from baseline to 12 weeks will be assessed. Physical activity will be quantified by measuring number of taken steps per day and will be measured using a validated wearable sensor named PAMSys. Monitoring of physical activity will be done during 48h baseline and 48 hour at 12 weeks.
Change in Quality of Life | Baseline and 12 weeks
  Quality of life will be assessed using a validated questionnaire, called PROMIS Global-10.
  The PROMIS Global-10 is a 10-item patient-reported questionnaire in which the response options are presented as 5-point (as well as a single 11-point) rating scales. The results of the questions are used to calculate two summary scores: a Global Physical Health Score and a Global Mental Health score. These scores are then standardized to the general population, using the "T-Score". The average "T-Score" for the United States population is 50 points, with a standard deviation of 10 points. Higher scores indicate a healthier patient.
change in depression | Baseline and 12 weeks
  Changes in depression from baseline to 12 weeks will be assessed. Depression will be quantified by the Center for Epidemiologic Studies Depression Scale (CES-D) at baseline and 12 weeks. The CES-D consists of 20 items, and each item is scored on a scale of 0 to 3, with 0 representing "Rarely or none of the time" and 3 representing "Most or all of the time." The total score for the CES-D ranges from 0 to 60, with higher scores indicating a greater severity of depressive symptoms.
  A score of 16 or higher is often considered as a cutoff point for identifying individuals who may be at risk for clinical depression. However, it is important to note that the CES-D is a screening tool, not a diagnostic tool, and a higher score should prompt further evaluation by a mental health professional.
Change in Fear of Falling | Baseline and 12 weeks
  Changes in Fear of falling will be assessed by Short Falls Efficacy Scale International (FES I) questionnaire at 12 weeks and will be compared to baseline measurements. Scores range from 16 to 64, the higher the score the more concerned the subject is with falling.
Change in Gait speed | Baseline and 12 weeks
  Change from baseline in Gait speed at 12 weeks. Gait speed will be measured using a validated wearable platform (LEGSys) during habitual walking speed.

OTHER OUTCOMES:
Supportive care acceptability | Baseline and 12 weeks
  To evaluate the acceptability of each in-home exercise program (both the tele-exergame and the non-tele-exergame exercises), we will employ a survey based on the Technology Acceptance Model. This survey will be administered to all participants, assessing their perceptions of ease of use, usefulness, technology anxiety, and intention to use.
  Each response will be rated on a 5-point Likert scale, ranging from "strongly disagree" to "strongly agree". This will be subsequently translated to a 0 to 4 scale for final evaluation, with higher scores indicating greater acceptability.
  The assessment will take place twice: initially at baseline, after the participants have tested the tele-exergame in the clinic for training purposes, and subsequently at the 12-week mark upon completion of the in-home exercise program.
Adherence | week 4, week 8, week 12
  We will assess adherence to the prescribed in-home exercise program through the use of an exercise diary and phone interview on monthly basis. In the intervention group (IG), we will also objectively quantify adherence. Adherence will be defined by the frequency and duration of in-home exercises performed over a 12-week period. We will record and review adherence data on a monthly basis for three months.
intervention related dropout | week 4, week 8, week 12
  We will categorize participants as intervention-related dropouts if they miss exercises for four consecutive weeks, decide to discontinue the exercise program, or experience any exercise-related adverse events. However, if a participant drops out due to non-exercise related reasons (e.g., developing a condition that limits their ability to participate in the program, passing away, traveling, relocating), we will not consider this an intervention-related dropout.
  Intervention-related dropout will be calculated as a percentage of the total number of participants in each group. We will collect this data on a monthly basis.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - UCLA, Los Angeles, California
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Park C, Mishra RK, York MK, Enriquez A, Lindsay A, Barchard G, Vaziri A, Najafi B. Tele-Medicine Based and Self-Administered Interactive Exercise Program (Tele-Exergame) to Improve Cognition in Older Adults with Mild Cognitive Impairment or Dementia: A Feasibility, Acceptability, and Proof-of-Concept Study. Int J Environ Res Public Health. 2022 Dec 6;19(23):16361. doi: 10.3390/ijerph192316361. PMID 36498431